CLINICAL TRIAL: NCT01197131
Title: Investigation of Urinary Steroid Metabolites in Children With Autism Spectrum Disorder
Brief Title: Urinary Steroid Metabolites in Autism
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Intersci Research Association, Austria (Other)
Responsible Party: Principal Investigator, Kurz Johann MD, Medical Doctor,, Intersci Research Association, Austria
Other Study IDs: protocol 1.0/18/06/2010
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: autism; autism spectrum disorder; steroids; steroid metabolites; urinary steroid metabolites; hormone formation; androgen precursor
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — noninvasive overnight urine (morning urine)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- autistic boys: Boys with autism spectrum disorder, age 5-15 years, diagnosis meets DSM-IV criteria ascertained by ADI-R or ADOS schedule or specialised paediatrician
- autistic girls: Girls with autism spectrum disorder, age 5-15 years, diagnosis meets DSM-IV criteria ascertained by ADI-R or ADOS schedule or specialised paediatrician.
- control boys: Healthy boys, age 5-15 years, mental status assessed by "Marburger Beurteilungsskala zum Asperger-Syndrome" (MBAS).
- control girls: Healthy girls, age 5-15 years, mental status assessed by "Marburger Beurteilungsskala zum Asperger Syndrome" (MBAS).

SUMMARY:
Deviation of hormone formation within nerve cells and nerve system provides autism spectrum disorder and neurodevelopment retardation through interaction of steroids with neurotransmitter-receptors, calcium-channel receptors and genomic interaction via nuclear steroid receptors.

Urinary steroid metabolites will be compared between children with autism spectrum disorder and healthy controls.

DETAILED DESCRIPTION:
Autism spectrum disorder presents many alterations in amino acid metabolism and in neurotransmitter systems (gamma amino acid system, glutamate-glutamine, nicotine-acid, serotonin-system) . Also alteration in gene activation within nerve cells and lymphocyte cultures encloses over 600 genes, affecting a wide field of enzymes , metabolic pathways and hormone formation. Male hormones and their precursors are often increased and their influence to nerve cell growth and spine formation is evident.

The diagnosis of autism spectrum disorder is made in accordance of criteria of the Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) of the American Psychiatric Association by an experienced and specialised paediatrician or psychologist and /or by an Autism Diagnostic Interview-Revised (ADI-R) or Autism Diagnostic Observation Schedule (ADOS) .

Overnight urine with measurement of quantity and time will be collected and a little part of the urinary samples will be frozen for storage till analysis. Age, weight and length of the children at collection time will be ascertained.

Four stratified groups (autistic boys, girls, and healthy controls, boys and girls, each age 5-15) will be formed.

Urinary samples will further remain anonymous through an Identification-Number (ID).

Analysis of hormones and the most of the known metabolites excreted in urine will be performed by a specialised laboratory using gas chromatography-mass spectrometry (GC/MS) analysis (University Hospital Bern, Steroid Laboratory, Switzerland).

The statistical analysis, with age, gender, weight, diagnosis and hormone analysis results as factors , consists in linear regression analysis to detect deviation in hormone formation and metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Autism spectrum disorder
* Age 5-15 years

Exclusion Criteria:

* Epilepsia
* Psychotropic medication
* other severe illness

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children , age 5-15 years with autism and autism spectrum disorder resident in Austria without other severe or psychiatric disorders.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
difference in hormone formation and androgen precursors | 3 years
  Calculation of hormone formation by comparison of urinary steroid metabolites

SECONDARY OUTCOMES:
difference in hormone formation in gender and age | 3 years
  Hormone formation depends on age and gender and will be calculated by comparison of urinary steroid metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Johann Kurz, MD, Principal Investigator — Intersci Research Association, Austria
Locations (1):
- Intersci Research Association, Leibnitz, Styria, Styria, Austria

REFERENCES:
- [Background] Hu VW, Nguyen A, Kim KS, Steinberg ME, Sarachana T, Scully MA, Soldin SJ, Luu T, Lee NH. Gene expression profiling of lymphoblasts from autistic and nonaffected sib pairs: altered pathways in neuronal development and steroid biosynthesis. PLoS One. 2009 Jun 3;4(6):e5775. doi: 10.1371/journal.pone.0005775. PMID 19492049
- [Background] Hu VW, Sarachana T, Kim KS, Nguyen A, Kulkarni S, Steinberg ME, Luu T, Lai Y, Lee NH. Gene expression profiling differentiates autism case-controls and phenotypic variants of autism spectrum disorders: evidence for circadian rhythm dysfunction in severe autism. Autism Res. 2009 Apr;2(2):78-97. doi: 10.1002/aur.73. PMID 19418574
- [Background] Purcell AE, Jeon OH, Zimmerman AW, Blue ME, Pevsner J. Postmortem brain abnormalities of the glutamate neurotransmitter system in autism. Neurology. 2001 Nov 13;57(9):1618-28. doi: 10.1212/wnl.57.9.1618. PMID 11706102
- [Background] Geier DA, Geier MR. A prospective assessment of androgen levels in patients with autistic spectrum disorders: biochemical underpinnings and suggested therapies. Neuro Endocrinol Lett. 2007 Oct;28(5):565-73. PMID 17984958
- See also: registration — http://www.controlled-trials.com/ISRCTN18725918/autism